CLINICAL TRIAL: NCT01398969
Title: A Prospective Randomized Multi-Centre Trial of Fresh vs. Frozen-and-Thawed FMT (Fecal Microbiota Transplantation) for Recurrent Clostridium Difficile Infection
Brief Title: Multi-Centre Trial of Fresh vs. Frozen-and-Thawed FMT for Recurrent CDI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Hamilton Health Sciences Corporation (Other); Kingston Health Sciences Centre (Other); Queen's University (Other); Vancouver General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDI.HBT.1
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2015-03

CONDITIONS: Clostridium Difficile Infection
Keywords: Randomized; Double Blind; Fecal Transplant; Recurrent; Clostridium difficile infection; CDI; HBT; Diarrhea; Frozen HBT; Thawed HBT; Fecal Enema
MeSH Terms: conditions — Clostridium Infections; Recurrence; Diarrhea | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Participants received either FMT or placebo to prevent further episode of CDI following FMT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh FMT (Experimental): Participants in this arm will receive Fresh FMT via rectal administration. They will be followed for 13 weeks to assess the cure or recurrence of CDI. All other procedures between the two arms will be identical.
  Interventions: Biological: Fresh FMT
- Frozen-and-Thawed FMT (Experimental): Participants in this arm will receive Frozen-and-Thawed FMT via rectal administration. They will be followed 13 weeks to assess the cure or recurrence of CDI. All other procedures between the two arms will be identical.
  Interventions: Biological: Frozen-and-Thawed FMT

INTERVENTIONS:
Biological: Fresh FMT — Participants will receive fresh FMT (supernatant of fecal specimen mixed with water) on day 1. If cure is not reached at day 5 (+3) a repeat FMT will be performed
  Other Names: Fresh Fecal Transplantation (FMT)
  Arms: Fresh FMT
Biological: Frozen-and-Thawed FMT — Participants will receive frozen-and-thawed FMT (supernatant of fecal specimen mixed with water) on day 1. If cure is not reached at day 5 (+3) a repeat FMT will be performed
  Other Names: Frozen-and-Thawed Fecal Transplantation (FMT)
  Arms: Frozen-and-Thawed FMT

SUMMARY:
The goal of this study is to determine the outcome of patients with recurrent CDI treated with fresh FMT versus frozen-and-thawed FMT in a randomized controlled trial. The specific objectives are to evaluate the safety of both types of FMT and to compare the clinical response, treatment failure and relapse rate in patients treated with fresh FMT compared to those treated with frozen-and-thawed FMT; also to assess the functional health and well-being of patients in each arm using a validated tool. The metagenomics will also be conducted from the stool samples collected from select patients from each arm: pre and post treatment and the matching donors. The metagenomics data will be used to determine the bacteria which may have contributed to the cure of CDI.

ELIGIBILITY:
Patient inclusion criteria

1. Age 18 years or older.
2. Able to provide informed consent.
3. Laboratory or pathology: confirmed diagnosis of recurrent CDI with symptoms (defined below) within the previous 180 days.
4. ≥ 2 episodes of CDI within 6 months and/or ongoing symptoms consistent with CDI despite treatment with oral vancomycin at a dose of at least 125 mg 4 times daily for at least 5 days.

Symptoms of CDI, diarrhea deﬁned as: 3 or more unformed bowel movements in 24 hours for a minimum of 2 days with no other causes for diarrhea. Subjects will be required to have laboratory or pathology-confirmed diagnosis of recurrent C. difficile infection where recurrence is deﬁned as return of diarrhea and positive stool test after a period of symptom resolution within 8 weeks of the first episode and has received at least a 10-day course of standard antibiotic therapy.

Patient exclusion criteria

1. Planned or actively participating in another clinical trial.
2. Patients with neutropenia with absolute neutrophil count <0.5 x 109/L
3. Evidence of toxic megacolon or gastrointestinal perforation on abdominal x-ray
4. Peripheral white blood cell count > 30.0 x 10E9/L AND temperature > 38.0 oC
5. Active gastroenteritis due to Salmonella, Shigella, E. coli 0157H7, Yersinia or Campylobacter.
6. Presence of colostomy
7. Unable to tolerate HBT or enema for any reason.
8. Requiring systemic antibiotic therapy for more than 7 days.
9. Actively taking Saccharomyces boulardii
10. Severe underlying disease such that the patient is not expected to survive for at least 30 days.
11. Any condition that, in the opinion of the investigator, that the treatment may pose a health risk to the subject.

Donor inclusion

1. Able to provide and sign informed consent.
2. Able to complete and sign the donor questionnaire
3. Able to adhere to fecal transplantation stool collection standard operating procedure.

Donor exclusion

1. Tested positive for any of the following: Human Immunodeficiency virus (HIV) 1/2, hepatitis IgM, hepatitis B (HBsAg), hepatitis C antibody, syphilis, human T- lymphotrophic virus (HTLV) 1/II and vancomycin resistant Enterococcus (VRE), methicillin resistant S. aureus (MRSA), Salmonella, Shigella, E.coli O157 H7, Yersinia and Campylobacter.
2. Detection of ova, parasites, C. difficile toxin, norovirus, adenovirus, rotavirus on stool examination
3. History of any type of active cancer or autoimmune disease
4. History of risk factors for acquisition of HIV, syphilis, Hepatitis B, Hepatitis C, prion or any neurological disease as determined by the donor questionnaire, appendix B.
5. History of gastrointestinal comorbidities, e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation or diarrhea
6. Receipt of blood transfusion from a country other than Canada in preceding 6 months
7. Antibiotic use or any systemic immunosuppressive agents in the 3 months prior to stool donation
8. Receipt of any type of live vaccine within 3 months prior to stool donation
9. Ingestion of nut or shell fish 3 days preceding donation if the recipient has known allergies to these food.
10. Any current or previous medical or psychosocial condition or behaviours which in the opinion of the investigator may pose risk to the recipients or the donor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The evaluation of the safety of HBT | 13 Weeks post HBT
  Assessment for adverse reactions in each study group by history, physical examination, blood work at baseline, day 12, week 5 and at completion (week 13) of the study period.
To determine the cure rate without recurrence of CDI at 13 weeks from the last HBT. | 13 Weeks post HBT

SECONDARY OUTCOMES:
To determine the relapse rate of clinical and laboratory evidence of CDI within the 13-week study period in participants treated with fresh HBT in comparison to frozen thawed HBT. | 13 Weeks post HBT
Assessment of the functional health and well-being of patients | Up to 1 year
  Patients will be asked to fill in the self-administered Health Survey at baseline, week 5, week 13 and 1 year from last HBT

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (4):
- Canada (4):
  - Vancouver Coastal Health (VCHRI/VCHA) - Diamond Health Care Centre and Vancouver General Hospital, Vancouver, British Columbia
  - St. Joseph's Hospital, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario

REFERENCES:
- [Derived] Lee CH, Steiner T, Petrof EO, Smieja M, Roscoe D, Nematallah A, Weese JS, Collins S, Moayyedi P, Crowther M, Ropeleski MJ, Jayaratne P, Higgins D, Li Y, Rau NV, Kim PT. Frozen vs Fresh Fecal Microbiota Transplantation and Clinical Resolution of Diarrhea in Patients With Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2016 Jan 12;315(2):142-9. doi: 10.1001/jama.2015.18098. PMID 26757463